CLINICAL TRIAL: NCT05704140
Title: Vienna Vascular Access Studied on Exchange of Dialysis Catheters for Shunts Where Feasible
Acronym: ViennaACTSNOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Austrian Society of Vascular Surgery (Unknown)
Responsible Party: Principal Investigator, Markus Plimon, MD, Head of the vascular access unit, Wilhelminenspital Vienna
Other Study IDs: 22-104-VK
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Haemodialysis; Dialysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- catheter based dialysis: All patients receiving catheter based dialysis in Vienna as of November 2022
  Interventions: Other: Catheter based Dialysis

INTERVENTIONS:
Other: Catheter based Dialysis — We will conduct a cross-section analysis regarding patients with catheter-based VA in Vienna.

SUMMARY:
We will conduct a cross-section analysis regarding patients with catheter-based vascular Access (VA) in Vienna.

Collected data will include demographic and clinical information such as age, gender, co-morbidities and imaging data from sonography and computer tomography.

Patients of interest will be assessed through a standardized clinician-executed questionnaire aimed at investigating their medical history regarding their VA.

Patients will be evaluated for the feasibility of an arteriovenous VA. Patients will receive standard of care ultrasound-based arterial and venous mapping.

DETAILED DESCRIPTION:
We will conduct a cross-section analysis regarding patients with catheter-based vascular Access (VA) in Vienna.

Collected data will include demographic and clinical information such as age, gender, co-morbidities and imaging data from sonography and computer tomography.

Patients of interest will be assessed through a standardized clinician-executed questionnaire aimed at investigating their medical history regarding their VA.

Patients will be evaluated for the feasibility of an arteriovenous VA. Patients will receive standard of care ultrasound-based arterial and venous mapping.

Study Rationale The rate of dialysis via catheter systems is around 40% in Vienna whereas in neighboring Germany this rate is historically below 15% according to the latest update of the Dialysis Outcomes and Practice Patterns Study. Therefore, possibly up to 20% of the patients receiving chronic dialysis in Vienna could be eligible for an arteriovenous VA. In absolute numbers we expect up to 400 patients.

By means of Vienna ACTS NOW the current situation will be meticulously assessed with the aim to improve the provision of medical care for dialysis patients in Vienna by exchanging catheters for arteriovenous VAs (where feasible and desired).

The collected data will serve as the basis of a future prospective interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and above
* Catheter-based dialysis as of 01.11.2022

Exclusion Criteria:

• Age lower than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving catheter based dialysis in Vienna at the specified timepoint
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Arteriovenous VA | December 2022-May 2023
  After a standard-of-care vascular mapping we will note the number of patients receiving catheter based dialysis who would be eligible for arteriovenous dialysis access.

SECONDARY OUTCOMES:
Reasons for catheter based dialysis | December 2022-May 2023
  We use a standardized questionnaire to assess the vascular access (VA) history of patients and why they are receiving catheter based dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Plimon, MD, Principal Investigator — Klinik Ottakring, Head of Departement of Vascular Surgery
Locations (1):
- Klinik Ottakring, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No